CLINICAL TRIAL: NCT07120191
Title: An Open Label Data Collection Study of My Connect Post-Op, a Post-Operative Communication Tool
Status: Recruiting | Type: Observational
Sponsor: Concentra AI, inc (Industry)
Responsible Party: Sponsor
Other Study IDs: CCAI-PostOp-2025-001
Record Dates: First submitted 2025-08-06; First posted 2025-08-13 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Total Hip Replacement; Total Knee Replacement
Keywords: Total joint replacement; post op communication; AI assisted conversation; artificial intelligence

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other

GROUPS / COHORTS (1):
- Adults undergoing total hip or knee replacement surgery: The entire active group will be utilizing the MyConnect Post Op communication tool.
  Interventions: Device: post op communication software

INTERVENTIONS:
Device: post op communication software — MyConnect Post Op is a communication tool that utilizes Technology Assisted Conversation to aid in the recovery of total knee and hip replacement patients
  Other Names: MyConnect Post Op

SUMMARY:
This open label, multi-center study will collect data from the participant's use of My Connect Post-Op Software as a post-operative communication solution in supporting patient recovery through Technology-Assisted Conversation (TAC). The application will be tested by patients who have undergone total joint replacement as a post-op communication tool. Data will be collected on how effectively the product guides patients through their recovery, identifying potential complications, and providing appropriate recommendations based on structured question pairs.

DETAILED DESCRIPTION:
Patients who are scheduled to undergo orthopedic total hip or total knee replacement surgery who meet the eligibility criteria will be enrolled in the study. Prior to surgery, participants will be trained on the use of the product and study requirements will be discussed. The training provides instructions at an in-office visit, outlining the device's usage. The instructions, along with warnings that the interface is with a computer and not a person, are emphasized in the device's app and user manual.

Daily prompts will interact with the patient, and the app will answer questions and direct specialized care/instructions. Participants will be instructed to engage with the software throughout the 30-day study period, responding to prompts and questions as the participant recovers from surgery. The software will log and archive all participants' interactions with the chatbot in the backend. Participants will be expected to utilize the investigational product after discharge and complete the 30-day study period.

For every active participant enrolled, a retrospective chart review patient from the same site will be enrolled in the study in a 1:1 manner. The retrospective review of approximately 200 patient's post-op clinical interactions will be collected as a control group for comparison.

An initial technical assessment of the application will be done with the first 10 active patients who have used the product for at least 2 weeks, focusing on the overall performance of the communication tool.

The primary objective of the study is to collect a structured conversation log, document product's decision-making patterns, and to ensure sufficient coverage of clinical scenarios.

Beyond the AI-driven conversation, the product will collect daily health characteristics on pain, sleep, activity levels, medication use, and diet. Pain reporting is captured through two distinct input methods: the GRASP® device, a trademarked handheld event marker used to record three distinct pain levels, and a smartphone-based slider, allowing for subjective pain self-reporting. The participant may choose either input method, both will be encouraged.

Additional product components include chat functionality and the provider dashboard.

Chat function will collect data for responsiveness, clarity, and patient engagement, ensuring it facilitates a smooth and intuitive post-operative communication experience. The provider dashboard will collect usability and functionality data, as it mirrors the patient's application while also allowing providers to manage office setup, input new patients, confirm surgical dates, and conduct real-time chat interactions with patients.

Both patient and provider satisfaction of the use of My Connect Post-Op Software will be collected periodically throughout the 30-day post-op period as noted in the Schedule of Activities.

ELIGIBILITY:
Inclusion Criteria:

Orthopedic patients scheduled for elective joint arthroplasty (single or double knee, or single or double hip replacement surgery).

Age 22-80 years. Owns a smart phone. Speaks and understands written and spoken English. Ability to give written informed consent.

Exclusion Criteria:

Known diagnosis of a psychiatric disorder. Known opioid dependence in the Investigator's opinion that may complicate participation.

Participation in another clinical trial investigating a drug, medical device, or a medical procedure in the 30 days preceding trial inclusion and throughout the duration of the trial.

Any condition that in the Investigator's opinion may complicate or preclude the subject from participating in this trial, such as physical impairment or noncooperation

Ages: 22 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: community sample from orthopedic practices
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2025-10-15 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Collect structured conversation logs | From enrollment to the end of treatment at 4 weeks
  Collect conversations between the participant and the clinically conversant AI

CONTACTS AND LOCATIONS:
Locations (1):
- Kansas Joint and Spine, Wichita, Kansas, United States

IPD SHARING:
Plan to Share IPD: Undecided